CLINICAL TRIAL: NCT00706511
Title: Sleep and Metabolism in Obesity: Impact of Gender
Brief Title: Metabolic Study of Sleep Apnea in Men and Women
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Chicago (Other)
Collaborators: Duke University (Other); Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 15870; P50HD057796 (NIH)
Record Dates: First submitted 2008-06-25; First posted 2008-06-27 (Estimated); Results first posted 2020-03-24 (Actual); Last update posted 2020-03-24 (Actual); Status verified 2016-09

CONDITIONS: Obstructive Sleep Apnea (OSA)
Keywords: OSA; Diabetes; Metabolism; Gender
MeSH Terms: conditions — Sleep Apnea, Obstructive; Diabetes Mellitus; Coitus

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Group with OSA (Experimental): Obese men and pre-menopausal women with OSA will receive 6 weeks of CPAP treatment, and assessed with a 3-day experimental protocol.
  Interventions: Device: CPAP
- Group without OSA (No Intervention): Obese men and pre-menopausal women without OSA will be characterized with a single 3-day experimental protocol

INTERVENTIONS:
Device: CPAP — CPAP (continuous positive airway pressure) treatment at home for 6 weeks
  Arms: Group with OSA

SUMMARY:
The purpose of this study is to look at the metabolic (use of energy) and hormonal features of sleep problems in men and women.

DETAILED DESCRIPTION:
Obesity is a major risk factor for obstructive sleep apnea (OSA), a condition characterized by repetitive respiratory disturbances, intermittent hypoxia, sleep fragmentation by frequent microarousals and low amounts of deep slow wave sleep (SWS). Today, more than 10 million American women suffer from OSA. OSA has been identified as an independent risk factor for the metabolic syndrome. Because OSA is more prevalent in men than in women, a disproportionate number of studies of OSA and its consequences have been conducted in men. Thus, OSA has been characterized as a disorder associated with gender-based health care inequity. Recent evidence, including data from our group, suggests that reduced amounts and intensity of SWS (i.e. slow-wave activity [SWA]) may play a pivotal role in the development of metabolic and cardiovascular disturbances in obese men and women, particularly those with OSA. This project will focus on sex differences in SWA and their relationship with daytime sleepiness and metabolic vulnerability in obese men and women with and without OSA. We propose to simultaneously characterize: 1. sleep-wake regulation; 2. measures of diabetes risk; 3. measures of cardiovascular risk; and 4. profiles of sex steroids, cortisol and adipokines in a. obese men without OSA, b. obese men with OSA before and after treatment with continuous positive airway pressure (CPAP), c. obese pre-menopausal women without OSA, and d. obese pre-menopausal women with OSA before and after CPAP treatment. The completion of these interdisciplinary studies will provide a unique data set contrasting in obese women versus obese men the relationships between sleep and the metabolic syndrome, OSA and the metabolic syndrome and the impact of CPAP treatment on the metabolic syndrome. This work will provide important insights regarding the pathophysiology of OSA and its adverse consequences in obese men and women, and the basis for the development of effective sex-specific prevention and treatment strategies.

ELIGIBILITY:
Inclusion Criteria:

* Obese (BMI of at least 30 kg/m2)

Exclusion Criteria:

* Clinically significant depression
* Positive pregnancy test
* Diagnosis of diabetes mellitus
* Hypertension (systolic > 140 mmHg and/or diastolic > 90 mmHg) not well-controlled on stable medication with either ACE inhibitors or diuretics
* Habitual alcohol use
* Excessive caffeine intake of more than 300 mg/day
* Hemoglobin < 11g/dL and/or hematocrit < 33%
* Systemic illnesses, including heart, renal, liver, or malignant disease
* Taking steroid preparations (including oral contraceptives), medications known to alter insulin secretion and/or action, or medications known to influence sleep during the 2 months prior to starting the study
* Travel across time zones during the 4 weeks prior to starting the study
* Irregular sleeping habits (including shift work)

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 27 (Actual)
Dates: Start 2007-12 (Actual); Primary Completion 2012-08-16 (Actual); Study Completion 2012-08-22 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Eve Van Cauter, Ph.D., Principal Investigator — University of Chicago
Locations (1):
- University of Chicago Department of Medicine, Section of Endocrinology, Diabetes & Metabolism, Chicago, Illinois, United States

REFERENCES:
- [Background] Tasali E, Leproult R, Ehrmann DA, Van Cauter E. Slow-wave sleep and the risk of type 2 diabetes in humans. Proc Natl Acad Sci U S A. 2008 Jan 22;105(3):1044-9. doi: 10.1073/pnas.0706446105. Epub 2008 Jan 2. PMID 18172212
- [Background] Tasali E, Van Cauter E, Ehrmann DA. Relationships between sleep disordered breathing and glucose metabolism in polycystic ovary syndrome. J Clin Endocrinol Metab. 2006 Jan;91(1):36-42. doi: 10.1210/jc.2005-1084. Epub 2005 Oct 11. PMID 16219719
- [Background] Tasali E, Mokhlesi B, Van Cauter E. Obstructive sleep apnea and type 2 diabetes: interacting epidemics. Chest. 2008 Feb;133(2):496-506. doi: 10.1378/chest.07-0828. PMID 18252916
- [Background] Knutson KL, Spiegel K, Penev P, Van Cauter E. The metabolic consequences of sleep deprivation. Sleep Med Rev. 2007 Jun;11(3):163-78. doi: 10.1016/j.smrv.2007.01.002. Epub 2007 Apr 17. PMID 17442599
- [Background] Van Cauter E, Holmback U, Knutson K, Leproult R, Miller A, Nedeltcheva A, Pannain S, Penev P, Tasali E, Spiegel K. Impact of sleep and sleep loss on neuroendocrine and metabolic function. Horm Res. 2007;67 Suppl 1:2-9. doi: 10.1159/000097543. Epub 2007 Feb 15. PMID 17308390
- [Background] Knutson KL, Ryden AM, Mander BA, Van Cauter E. Role of sleep duration and quality in the risk and severity of type 2 diabetes mellitus. Arch Intern Med. 2006 Sep 18;166(16):1768-74. doi: 10.1001/archinte.166.16.1768. PMID 16983057
- [Background] Latta F, Leproult R, Tasali E, Hofmann E, L'Hermite-Baleriaux M, Copinschi G, Van Cauter E. Sex differences in nocturnal growth hormone and prolactin secretion in healthy older adults: relationships with sleep EEG variables. Sleep. 2005 Dec;28(12):1519-24. doi: 10.1093/sleep/28.12.1519. PMID 16408410
- See also: University of Chicago Sleep Disorders Center — http://www.uchospitals.edu/specialties/pulmonary/sleep-disorders/index.html

RESULTS

PARTICIPANT FLOW:
Groups:
- Men With OSA; Women With OSA: Obese men and pre-menopausal women with OSA will receive 6 weeks of CPAP treatment, and assessed with a 3-day experimental protocol.
  CPAP: CPAP (continuous positive airway pressure) treatment at home for 6 weeks
- Men Without OSA; Women Without OSA: Obese men and pre-menopausal women without OSA will be characterized with a single 3-day experimental protocol
Period: Overall Study
Arm/Group | Men With OSA | Women With OSA | Men Without OSA | Women Without OSA
Started | 10 | 4 | 3 | 10
Completed | 9 | 4 | 3 | 10
Not Completed | 1 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 1 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Men With OSA | Women With OSA | Men Without OSA | Women Without OSA | Total
Number analyzed (Participants) | 10 | 4 | 3 | 10 | 27
Age, Continuous [Mean (Standard Deviation); unit: years] | 37.7 (6.5) | 35 (2.9) | 24.7 (1.5) | 31.9 (7.4) | 33.7 (7.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 4 | 0 | 10 | 14
  Male | 10 | 0 | 3 | 0 | 13
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
  Black or African American | 2 | 4 | 2 | 7 | 15
  White | 8 | 0 | 1 | 3 | 12
  More than one race | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Polysomnography - Apnea-hypopnea Index (AHI)
Description: apnea-hypopnea index: number of apneas and hypopneas per hour of recording; a measure of the severity of obstructive sleep apnea; varies from min=0 to max=120; AHI between 0 and <5: no significant sleep apnea; AHI between 5 and <15: mild sleep apnea; AHI between 15 and <30: moderate sleep apnea; AHI of 30 and above: severe sleep apnea.
Time Frame: After 6 weeks of CPAP (Treatment)
Population: One participant (a men with OSA) was excluded in the analysis because he did not complete the study. (See the participant flow chart)
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Men With OSA | Women With OSA | Men Without OSA | Women Without OSA
Number analyzed (Participants) | 9 | 4 | 3 | 10
units on a scale | 11.4 (13.7) | 0.7 (0.8) | 6 (5.2) | 1.1 (1.5)

2. Primary Outcome: Polysomnography - Minutes of N3 Stage
Description: Stage N3, sometimes referred to as "delta sleep" or "slow wave sleep", is characterized by slow waves in the electro-encephalogram (EEG) that reflect synchronization of firing of cortical neurons. N3 sleep is considered the most restorative stage of sleep for both the brain and the rest of the body.
Time Frame: After 6 weeks of CPAP (Treatment)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: minutes
Arm/Group | Men With OSA | Women With OSA | Men Without OSA | Women Without OSA
Number analyzed (Participants) | 9 | 4 | 3 | 10
minutes | 58.1 (42.6) | 53.7 (28.7) | 75.7 (22.4) | 66.6 (30.6)

3. Primary Outcome: Polysomnography - Minutes of REM Stage
Time Frame: After 6 weeks of CPAP (Treatment)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: minutes
Arm/Group | Men With OSA | Women With OSA | Men Without OSA | Women Without OSA
Number analyzed (Participants) | 9 | 4 | 3 | 10
minutes | 98.2 (24.1) | 101.5 (10.9) | 107.8 (28.2) | 111.1 (24.1)

4. Primary Outcome: Polysomnography - Sleep Efficiency
Description: Sleep efficiency: a measure of objective sleep quality; calculated from the polygraphic sleep recording as the ratio of time spent asleep during the scheduled sleep period to total scheduled sleep period. Expressed in %. Varies from 0% (the subject did not sleep at all) to 100% (the subject spent the entire scheduled sleep period asleep).
Time Frame: After 6 weeks of CPAP (Treatment)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Men With OSA | Women With OSA | Men Without OSA | Women Without OSA
Number analyzed (Participants) | 9 | 4 | 3 | 10
score on a scale | 88.9 (6.2) | 89.9 (6.5) | 86.5 (6.3) | 89.7 (5)

5. Secondary Outcome: IVGTT (Intravenous Tolerance Test) - Sensitivity Index (SI)
Description: Sensitivity Index (SI): a measure of how much insulin the body needs to metabolize a given amount of glucose. SI is calculated using a mathematical model describing the profiles of blood glucose and serum insulin after intravenous glucose injection. SI varies from 0 to an undefined upper limit but generally under 20. Higher values of SI represent a better outcome.
Time Frame: After treatment (6 weeks)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Men With OSA | Women With OSA | Men Without OSA | Women Without OSA
Number analyzed (Participants) | 9 | 4 | 3 | 10
score on a scale | 1.226 (0.642) | 1.106 (0.44) | 2.32 (1.15) | 4.195 (3.346)

6. Secondary Outcome: IVGTT (Intravenous Tolerance Test) - Acute Insulin Response
Description: Acute Insulin Response is calculated as the area under the insulin curve for the first 19 minutes after intravenous glucose injection. "Area under the insulin curve" is expressed in pmol x min/L.
Time Frame: After treatment (6 weeks)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: pmol x min/L
Arm/Group | Men With OSA | Women With OSA | Men Without OSA | Women Without OSA
Number analyzed (Participants) | 9 | 4 | 3 | 10
pmol x min/L | 1061 (736) | 623 (338) | 734 (784) | 1020 (564)

7. Secondary Outcome: IVGTT (Intravenous Tolerance Test) - Disposition Index (DI)
Description: Disposition Index (DI) is the product of sensitivity index (SI) by the amount of insulin secreted in response to blood glucose levels. It is a marker of the risk of type 2 diabetes. Low DI reflects a high risk of diabetes. DI can vary from 0 to an undefined upper limit. The physiological range for the Disposition Index is 500 to 5,000. Higher values represent a better outcome.
Time Frame: After treatment (6 weeks)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Men With OSA | Women With OSA | Men Without OSA | Women Without OSA
Number analyzed (Participants) | 9 | 4 | 3 | 10
score on a scale | 1159 (789) | 683 (531) | 1257 (849) | 3718 (3270)

ADVERSE EVENTS:
Time Frame: Up to 24 hours
Arm/Group | Group With OSA | Group Without OSA
All-Cause Mortality (participants affected / at risk) | 0/13 | 0/13
Serious Adverse Events (participants affected / at risk) | 0/13 | 0/13
Other Adverse Events (participants affected / at risk) | 0/13 | 0/13

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No